CLINICAL TRIAL: NCT04380532
Title: Clinical Trial of COVID-19 Therapeutic Vaccine Formulated as an Oral Pill
Brief Title: Tableted COVID-19 Therapeutic Vaccine
Acronym: COVID-19
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Immunitor LLC (Industry)
Collaborators: Immunitor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Imm24
Record Dates: First submitted 2020-04-29; First posted 2020-05-08 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Covid19
Keywords: COVID-19; SARS-CoV-2; coronavirus; respiratory disease; SARS; ARDS; pneumonia; pandemic
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Respiration Disorders; Pneumonia

STUDY DESIGN:
Intervention Model Description: Healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V-SARS recipients (Experimental): Single arm having at least 20 volunteers administered once-per-day pill of V-SARS
  Interventions: Biological: V-SARS

INTERVENTIONS:
Biological: V-SARS — Therapeutic vaccine formulated as a pill derived from heat-inactivated plasma from COVID-19 patients administered once-per-day to at least 20 healthy volunters for at least one month

SUMMARY:
Safety and immunogenicity one-month study in healthy individuals administered once-daily pill of therapeutic vaccine made from heat-inactivated plasma from donors with COVID-19. Healthy, at least 20, volunteers will be monitored for signs of adverse events. Their PBMC will be collected at baseline and one month later to analyze which type of immune response vaccine has induced.

DETAILED DESCRIPTION:
Experimental batch of tableted thermostable vaccine obtained from pooled plasma of COVID-19 patients is produced. The goal of this trial is test safety and immunogenicity of once-per-day day administered orally to volunteers for 15 days. Baseline and post-treatment standard safety parameters will be compared. Blood samples from volunteers will be monitored and immunogenicity lab assays will be undertaken to characterize immune response.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cases of Covid-19 (all by RT-PCR from same laboratory)
* Mild to severe clinical presentation (identified at the time of admission to ward by National Early Warning Score NEWS-2; mild 0-4; severe 5-6)

Exclusion Criteria:

* Unable to take oral medication,
* Immunocompromised
* Known comorbid condition like hypertension, cardiovascular disease, diabetes mellites, asthma, COPD, cerebrovascular disorder, malignancy of any type, pregnancy,
* BMI less than 18
* Smoking history (more than one pack per day)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Effect on CBC as per CTCAE v4.0 | 15 Days
  Routine laboratory complete blood cell count at pre- and post-treatment periods by automated CBC counter Routine laboratory complete blood count Routine clinical laboratory CBC parameters at pre- and post-treatment periods
Effect on biochemistry parameters as per CTCAE v4.0 | 15 Days
  Routine clinical laboratory blood biochemistry parameters at pre- and post-treatment periods by automated biochemistry analyzer

SECONDARY OUTCOMES:
Lack of adverse events as per CTCAE v4.0 | 15 days
  Clinical well-being assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Aldar Bourinbayar, MD/PhD, Principal Investigator — Immunitor LLC
Locations (2):
- Immunitor Inc, Vancouver, BC - British Columbia, Canada
- Aldar Bourinbayar, Ulaanbaatar, BZD, 3-khoroo, Mongolia

IPD SHARING:
Plan to Share IPD: Yes
Free dissemination of published data
Supporting Information: Study Protocol
Time Frame: when become public
Access Criteria: non-confidential data
URL: http://immunitor.com

REFERENCES:
- [Background] Silin DS, Lyubomska OV, Jirathitikal V, Bourinbaiar AS. Oral vaccination: where we are? Expert Opin Drug Deliv. 2007 Jul;4(4):323-40. doi: 10.1517/17425247.4.4.323. PMID 17683247